CLINICAL TRIAL: NCT06989541
Title: Immunoglobulin for Hypogammaglobulinemia Due to Chimeric Antigen Receptor T Cell Therapy
Acronym: ICART
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-24-0422
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hypogammaglobulinemia, Acquired
Keywords: secondary immunodeficiency; CAR T; immune globulin
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVIG: Intravenous Immunoglobulin Replacement
  Interventions: Biological: Immune Globulin Intravenous (Human), 10%
- SCIG: Subcutaneous Immunoglobulin Replacement
  Interventions: Biological: Immune Globulin Subcutaneous (Human), 20% Solution

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10% — Intravenous immune globulin replacement
  Groups: IVIG
Biological: Immune Globulin Subcutaneous (Human), 20% Solution — Subcutaneous immune globulin replacement
  Groups: SCIG

SUMMARY:
Chimeric antigen receptor (CAR) T cells are special immune cells taken from a patient and changed in a lab to help them find and attack cancer cells. These cells are designed to look for a marker called CD19, which is found on both cancer cells and healthy B cells (a type of white blood cell). Because of this, CAR T cells can also destroy healthy B cells. This can lead to a strong drop in B cells and cause a condition called hypogammaglobulinemia (HGG), which makes it harder for the body to fight infections. Serious infections are common in people treated with CAR T cells and are a major reason for death that is not caused by the return of cancer.

To help prevent infections, patients with HGG often get immunoglobulin replacement therapy (IRT), which gives them the antibodies they need. This treatment can be given through a vein (IVIG) or under the skin (SCIG). The goal of this project is to study how often these patients get bacterial infections, how they feel about their quality of life and treatment, and what side effects they may have when treated with IVIG or SCIG after CAR T-cell therapy.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cells are patient-derived T cells engineered to express a fusion protein that directs them to target a tumor-associated antigen. The tumor-associated antigen CD19 is expressed on tumor cells in these conditions as well as on healthy cells of the B cell lineage. This results the "on-target off-tumor" effect of profound B cell depletion in these patients often with attendant hypogammaglobulinemia (HGG). Serious infections are common in this patient population and represent the main cause of non-relapse related mortality in CAR T cell treated patients.

Treatment of HGG with immunoglobulin replacement therapy (IRT) is a core component of infection prevention. Standard of care IRT can be administered intravenously (IVIG) or subcutaneously (SCIG). The proposed project will investigate frequency of bacterial infections, quality of life, treatment satisfaction, and adverse events in patients treated with CAR T-cell therapy who are treated with IVIG and SCIG.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Severe HGG defined as total IgG <4 g/L (after subtracting the IgG paraprotein fraction, if present)
3. Treated with CD19 targeted CAR T cell therapy in the past 6 months
4. Consent to receive plasma-derived productions
5. Ability to provide informed consent

Exclusion Criteria:

1. Inability to comply with study procedures
2. Pregnancy or planning to conceive
3. Breastfeeding
4. Protein-losing conditions that may contribute to HGG (e.g., protein-losing enteropathy, nephrotic syndrome)
5. SCIG infusion in the prior 3 months.
6. History of allergy or severe reactions to immune globulin productions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with CD19 targeted CAR T cell therapy for B cell malignancy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Time normalized rate of infections grade 3 or greater | 40 weeks
  Time normalized rate of infections grade 3 or greater

SECONDARY OUTCOMES:
Time normalized rate of validated infections | 40 weeks
  Time normalized rate of infections (per subject-year) confirmed using microbiologic, clinical, and radiologic criteria
Days on therapeutic antibiotics | 40 weeks
  Days on therapeutic antibiotics for treatment of an infection (excluding days on routinely provided prophylactic antibiotics)
Days missed work/school/unable to perform normal daily activities due to infections | 40 weeks
  Days missed work/school/unable to perform normal daily activities due to infections (rate per subject-year)
Total number of days of hospitalizations due to infections | 40 weeks
  Total number of days of hospitalizations due to infections (rate per subject-year)
Geometric mean of IgG serum trough concentration | 40 weeks
  Geometric mean of IgG serum trough concentration at last study visit
Mean TSQM9 | 40 weeks
  Treatment Satisfaction Questionnaire for Medication (TSQM9)
IRT-related adverse events | 40 weeks
  Nature and frequency of immune globulin-related adverse events
Hours of infusion clinic time required for IVIG administration | 40 weeks
  Hours of infusion clinic time required for IVIG administration
Mean total grams of immunoglobulin administered | 40 weeks
  Mean total grams of immunoglobulin administered per patient-year
Mean leukocyte counts at the last study visit | 40 weeks
  Mean leukocyte counts at the last study visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No